CLINICAL TRIAL: NCT07235176
Title: A Phase Ib/II Clinical Study to Evaluate Safety, Preliminary Efficacy and PK Characteristic of QLS1304 Combined With Endocrine Therapy in ER+/HER2- Breast Cancer Patients
Brief Title: Phase Ib/II Clinical Study of QLS1304 Combined With Endocrine Therapy in the Treatment of ER+/HER2- Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS1304-201
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced ER+/HER2- Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLS1304 tablet + SERD (Experimental)
  Interventions: Drug: QLS1304 tablet+Fulvestrant or QLC1401
- QLS1304 tablet + ET+CDK4/6i (Experimental)
  Interventions: Drug: QLS1304 tablet+Fulvestrant，AI or QLC1401+CDK4/6i

INTERVENTIONS:
Drug: QLS1304 tablet+Fulvestrant or QLC1401 — QLS1304 combined with endocrine therapy
  Arms: QLS1304 tablet + SERD
Drug: QLS1304 tablet+Fulvestrant，AI or QLC1401+CDK4/6i — QLS1304 combined with endocrine therapy
  Arms: QLS1304 tablet + ET+CDK4/6i

SUMMARY:
This study is a multi-center, open label, phase Ib/II clinical trial aimed at evaluating the safety, preliminary efficacy characteristic and PK characteristics of QLS1304 in combined with endocrine therapy in ER+/HER2- breast cancer patients. This study was divided into two stages: combo dose escalation and dose expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study, sign an informed consent form and have good compliance;
2. Age ≥ 18 years old, Male or female
3. ECOG score: 0-1
4. Expected survival ≥ 12 weeks
5. Local recurrent or metastatic advanced ER+/HER2- breast cancer confirmed by histopathology or cytopathology;
6. Failed to at least one therapy line of endocrine therapy ;
7. Baseline presence of at least one measurable lesion according to the RECIST v1.1;
8. The functional level of important organs is basically normal, meeting the requirements of the scheme;
9. Female subjects with fertility and male subjects must agree to use highly effective contraception during the study treatment period and within 180 days after the last medication;
10. Female subjects with fertility must have a negative serum HCG test within 7 days before the first medication in the study, and must be in non lactation.
11. Volunteer to participate in this clinical trial, willing and able to follow the procedures related to clinical visits and research, understand the research procedures, and have signed informed consent.

Exclusion Criteria:

1. Subjects have received live or attenuated live vaccines within 4 weeks before the first use of the investigational drug.
2. Subjects have undergone major organ surgery within 4 weeks before the first use of the investigational drug.
3. Subjects require long-term or high-dose use of non-steroidal drugs.
4. Subjects have not recovered from adverse events (AEs) caused by previous anti-tumor treatment to ≤ grade 1.
5. Subjects have a known or suspected severe allergy to the investigational drug or any of its components.
6. Subjects have other active malignant tumors within 5 years before the first use of the investigational drug.
7. Subjects have brain metastases and/or carcinomatous meningitis or leptomeningeal disease.
8. Subjects have active tuberculosis, radiation pneumonitis, drug-induced pneumonitis, pulmonary fibrosis, or other diseases, symptoms, or signs of severe lung function impairment.
9. Subjects are unable to swallow tablets or had gastrointestinal abnormalities that the investigator assessed as potentially affecting drug absorption.
10. Subjects have a history of severe cardiovascular or cerebrovascular disease within 6 months before the first use of the investigational drug.
11. Subjects have a hypertension medial history that blood is not well controlled despite treatment with multiple antihypertension drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-11-02 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) of QLS1304 in combo therapy | through study completion，an average of 2 years
objective response rate（ORR） | through study completion，an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China